CLINICAL TRIAL: NCT04214132
Title: Evaluation of a Virtual Counseling Application for Communication Skills Training in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Shefaly Shorey, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NUS S-18-074
Record Dates: First submitted 2019-12-22; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Communication
Keywords: Virtual reality; Learning; Technology; Patients
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual patients group (Experimental): Only nursing undergraduates from AY2017/2018 cohort, who have completed the redesigned NUR1110 (Effective Communication for Health-Professionals) core module will receive additional training using Virtual Patients in each semester (2 semesters per year) of year 2 and year 3 before they go for the clinical posting. Students will have unlimited access to the Virtual Patients (available scenarios depend on which semester the student is in) by logging in through the school portal.
  Interventions: Other: Virtual Counselling Application using Artificial Intelligence
- Blended learning group (No Intervention): Nursing undergraduates from AY2016/2017 cohort who who have completed the redesigned NUR1110 (Effective Communication for Health-Professionals) core module that comprised of weekly online e-lectures and face-to-face tutorials.

INTERVENTIONS:
Other: Virtual Counselling Application using Artificial Intelligence — Intervention comprises of four Virtual Patients scenarios that aimed to improve nursing undergraduates communication skills in a clinical setting. These scenarios are based on authentic clinical cases (adapted from the real-life clinical case studies) focusing mainly on the communication aspects. Scenarios included 1) a middle-aged pregnant woman in her third trimester experiencing pain, 2) a middle-aged lorry driver who self-admitted to the hospital due to relapse of depressive symptoms, 3) changing a bloody dressing of a middle-aged male patient who had an operation 3 days ago, and 4) communicating with a fellow stressed student during their final preregistration clinical posting period.
  Arms: virtual patients group

SUMMARY:
The Alice Lee Centre for Nursing Studies under the National University of Singapore offers a three-years (four years for honors students), full-time Bachelor of Science (Nursing) program that is accredited by the Singapore Nursing Board. The course covers core modules such as, anatomy, physiology and physical assessment, pathophysiology, pharmacology and nursing practice, communication and cultural diversity, and includes clinical practicums at tertiary hospitals that range from two weeks to three months.

This project will be carried out with nursing undergraduates of National University of Singapore who had completed the core module NUR1110 (Effective Communication for Health Professionals) in their year 1 of nursing courses. The 2-year study will follow these students in year 2 and year 3 consecutively by introducing Virtual Patients (VP) depicting real-life case scenarios at gradual difficulty levels before their end-of-semester clinical posting. Four VP case scenarios were developed for each semester on the following topics: 1) interview a pregnant woman with pain to solicit holistic history taking (year 2 semester 1); 2) history taking from a depressed patient (year 2 semester 2); 3) use of a standardized approach such as Situation, Background, Assessment, and Recommendation (SBAR) to hand off interdisciplinary communications (year 3 semester 1); and 4) showing empathy to the fellow nursing student (year 3 semester 2).

Overall, the aim of this project is to develop and evaluate the use of VPs in better preparing nursing undergraduates in communicating with real-life patients, family members, and other healthcare professionals during their clinical posting. The specific research questions the investigators plan to answer in this project are as follows:

1. What is the effect of using VPs in enhancing nursing undergraduates' self-efficacy and attitude toward learning communication skills?
2. Do the students receiving additional training using VPs perform better in their communication skills during the clinical posting compared with students receiving standard training?
3. What are the levels of outcomes of students' self-efficacy and attitude toward learning communication skills at pretest (semester 1, year 2 before receiving the VP training), posttest 1 (last day of clinical posting year 2 semester 1), posttest 2 (last day of clinical posting year 2 semester 2), posttest 3 (last day of clinical posting year 3 semester 1), and posttest 4 (last day of clinical posting year 3 semester 2)?
4. What are the changes in self-efficacy and attitude toward communication skills scores over time (pretest, posttests 1-4)?
5. What are the students' experiences in receiving additional training using VPs before their clinical posting? The aim of this paper is therefore to provide a detailed breakdown on the development process of the Virtual Counseling Application using Artificial Intelligence (VCAAI) for communication skills training in nursing education and to highlight challenges faced and recommended resolutions to inform future research.

ELIGIBILITY:
Inclusion Criteria:

* Year two nursing undergraduates
* Enrolled for Bachelor of Science (Nursing) course for Academic years 2017/2018 at Alice Lee Center for Nursing Studies, NUS.
* Completed the core module "Effective Communication for Health Professionals" in Year 1
* Able to read and speak English fluently

Exclusion Criteria:

* Medical or mental illness that may hinder the use of Virtual Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Mean score of students' attitude towards learning communication skills | at 4 months
  Measured using a self-report, 26-items Communication Skills Attitude Scale (CSAS) that uses a 5-point Likert scale (1=strongly disagree, 5=strongly agree), and has a total score of 130. A higher score indicate more positive attitude towards learning communication skills. Within cohort comparison.
Mean score of students' attitude towards learning communication skills | at 12 months
  Measured using a self-report, 26-items Communication Skills Attitude Scale (CSAS) that uses a 5-point Likert scale (1=strongly disagree, 5=strongly agree), and has a total score of 130. A higher score indicate more positive attitude towards learning communication skills. Within cohort comparison.
Mean score of students' attitude towards learning communication skills | at 16 months
  Measured using a self-report, 26-items Communication Skills Attitude Scale (CSAS) that uses a 5-point Likert scale (1=strongly disagree, 5=strongly agree), and has a total score of 130. A higher score indicate more positive attitude towards learning communication skills. Within cohort comparison.
Mean score of students' attitude towards learning communication skills | at 24 months
  Measured using a self-report, 26-items Communication Skills Attitude Scale (CSAS) that uses a 5-point Likert scale (1=strongly disagree, 5=strongly agree), and has a total score of 130. A higher score indicate more positive attitude towards learning communication skills. Within cohort comparison.
Mean score of students' perceived self-efficacy | at 4 months
  Communication skills sub-scale of the Nursing students self-efficacy scale. 8-items using a 5-point likert scale (0=not at all confident, 5= completely confident) with a total score of 40. A higher score indicates a higher perceived communication self-efficacy. Within cohort comparison.
Mean score of students' perceived self-efficacy | at 12 months
  Communication skills sub-scale of the Nursing students self-efficacy scale. 8-items using a 5-point likert scale (0=not at all confident, 5= completely confident) with a total score of 40. A higher score indicates a higher perceived communication self-efficacy. Within cohort comparison.
Mean score of students' perceived self-efficacy | at 16 months
  Communication skills sub-scale of the Nursing students self-efficacy scale. 8-items using a 5-point likert scale (0=not at all confident, 5= completely confident) with a total score of 40. A higher score indicates a higher perceived communication self-efficacy. Within cohort comparison.
Mean score of students' perceived self-efficacy | at 24 months
  Communication skills sub-scale of the Nursing students self-efficacy scale. 8-items using a 5-point likert scale (0=not at all confident, 5= completely confident) with a total score of 40. A higher score indicates a higher perceived communication self-efficacy. Within cohort comparison.

SECONDARY OUTCOMES:
clinical communication skills mean scores | 4 months (after completion of Year 2 semester 1 clinical posting)
  Clinical assessment scores by clinical instructors obtained through the online clinical management system. Performance scores will be compared with the previous cohort that did not have virtual patient training.
  The Entrustable Professional Activities (EPA) assessment scale comprises of 7-items, each with a score of 1 to 5, and a total score of 35. The higher the score the better the communication performance.
clinical communication skills mean scores | 12 months (after completion of Year 2 semester 2 clinical posting)
  Clinical assessment scores by clinical instructors obtained through the online clinical management system. Performance scores will be compared with the previous cohort that did not have virtual patient training.
  The Entrustable Professional Activities (EPA) assessment scale comprises of 7-items, each with a score of 1 to 5, and a total score of 35. The higher the score the better the communication performance.
clinical communication skills scores | 16 months (after completion of Year 3 semester 1 clinical posting)
  Clinical assessment scores by clinical instructors obtained through the online clinical management system. Performance scores will be compared with the previous cohort that did not have virtual patient training.
  The Entrustable Professional Activities (EPA) assessment scale comprises of 7-items, each with a score of 1 to 5, and a total score of 35. The higher the score the better the communication performance.
clinical communication skills scores | 24 months (after completion of Year 3 semester 2 clinical posting)
  Clinical assessment scores by clinical instructors obtained through the online clinical management system. Performance scores will be compared with the previous cohort that did not have virtual patient training.
  The Entrustable Professional Activities (EPA) assessment scale comprises of 7-items, each with a score of 1 to 5, and a total score of 35. The higher the score the better the communication performance.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No